CLINICAL TRIAL: NCT00942253
Title: The Effects of Exercise Training in Combination With Dopamine Agonist to Physical Fitness Parameters and Quality of Life in Dialysis Patients With the Restless Legs Syndrome.
Brief Title: Exercise Training in Dialysis Patients With Restless Legs Syndrome (RLS)
Acronym: HDRLS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Thessaly (Other)
Collaborators: Center for Research and Technology Thessaly - CERETETH (Unknown); European Social Fund (Other)
Responsible Party: Dr. Giorgos K. Sakkas, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 3745/EPE/2006; 04EP-07/8.3/04EP-Greece
Record Dates: First submitted 2009-07-17; First posted 2009-07-20 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-07

CONDITIONS: Restless Legs Syndrome; End Stage Renal Disease; Hemodialysis; Muscle Cachexia; Sleep Disorders
Keywords: RLS; Muscle; Dialysis; exercise; dopamine agonist; Sleep
MeSH Terms: conditions — Restless Legs Syndrome; Kidney Failure, Chronic; Sleep Wake Disorders; Motor Activity | interventions — Dopamine Agonists; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dopamine Agonist Group (Experimental): Dialysis patients will receive dopamine agonist for 24 weeks following a 24 weeks period of combined treatment with dopamine agonist and aerobic intradialytic exercise.
  Patients will be given evening doses of dopamine agonists, 2 hours before bedtime. The dopamine agonists' dose will be 0.25 mg/dose and remain constant until the end of the study.
  Interventions: Other: Dopamine Agonist and Exercise
- Placebo Group (Placebo Comparator): Dialysis patients will receive placebo for 24 weeks following a 24 weeks period of combined treatment with placebo and aerobic intradialytic exercise.
  Patients will be given evening doses of placebo, 2 hours before bedtime.
  Interventions: Other: Dopamine Agonist and Exercise

INTERVENTIONS:
Other: Dopamine Agonist and Exercise — Dialysis patients will receive dopamine agonist or placebo for 24 weeks following a 24 weeks period of combined treatment with dopamine agonist or placebo and aerobic intradialytic exercise.

SUMMARY:
Uremic etiology Restless legs syndrome (RLS) has been associated with poorer quality of life (QoL) compared to RLS-free counterparts mainly due to sleep deprivation factors. Exercise training in hemodialysis (HD) patients with RLS has been proven to be a safe approach in temporally ameliorating RLS symptoms similarly to the use of pharmacological treatment with dopamine agonists. However it not known whether the exercise anabolic stimulus and the dopamine agonist treatment could act synergistically for the improvement of physical functioning and muscle performance as well as in the amelioration of augmentation symptoms in hemodialysis patients with RLS.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled study to evaluate the acute and long term (6 months) effect of exercise training in combination with dopamine agonists in quality of life, muscle function, sleep quality and metabolism in patients with restless legs syndrome (RLS) receiving dialysis therapy.

Objectives - Aims:

1. To investigate whether a single bout of intradialytic exercise session could have an effect in motor restlessness often seen during hemodialysis session in patients with RLS
2. To investigate whether a 24 weeks therapy with dopamine agonist or placebo will have an effect in sleep quality, functional capacity and metabolic profile of the hemodialysis patients with RLS
3. To examine whether dopamine agonists or placebo and aerobic intradialytic exercise act synergistically for the improvement of physical functioning and muscle performance as well as it could reduce the signs of augmentation in hemodialysis patients with RLS

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable hemodialysis patients with positive diagnosis in IRLSS questionnaire for the RLS will be eligible to participate. Entry criteria included being on chronic hemodialysis for six months, able to perform an exercise training, with dialysis delivery (KT/V) > 1.1.

Exclusion Criteria:

* Patients were excluded from the study if they were diagnosed with neuropathies or reasons for being in a catabolic state (including malignancies, HIV and opportunistic infections, active inflammation), within 3 months prior to the start of the study. In addition patients treated with drugs recommended for the treatment of RLS as well as patients with Parkinson's disease or untreated depression will be also excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2006-09; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
IRLS severity scale | 24 and 48 wks

SECONDARY OUTCOMES:
Quality of Life Quality of Sleep Functional Capacity Muscle Size and composition Body Composition Glucose Tolerance Heart and respiratory functionality | 24 and 48 wks

CONTACTS AND LOCATIONS:
Overall Officials: Giorgos K Sakkas, PhD, Principal Investigator — UTH - CERETETH; Ioannis Stefanidis, MD PhD, Study Chair — UTH
Locations (1):
- University Hospital of Larissa, Nephrology Clinic, Larissa, Thessaly, Greece

REFERENCES:
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639
- [Derived] Giannaki CD, Sakkas GK, Karatzaferi C, Maridaki MD, Koutedakis Y, Hadjigeorgiou GM, Stefanidis I. Combination of Exercise Training and Dopamine Agonists in Patients with RLS on Dialysis: A Randomized, Double-Blind Placebo-Controlled Study. ASAIO J. 2015 Nov-Dec;61(6):738-41. doi: 10.1097/MAT.0000000000000271. PMID 26262586
- [Derived] Giannaki CD, Sakkas GK, Karatzaferi C, Hadjigeorgiou GM, Lavdas E, Kyriakides T, Koutedakis Y, Stefanidis I. Effect of exercise training and dopamine agonists in patients with uremic restless legs syndrome: a six-month randomized, partially double-blind, placebo-controlled comparative study. BMC Nephrol. 2013 Sep 11;14:194. doi: 10.1186/1471-2369-14-194. PMID 24024727
- [Derived] Giannaki CD, Hadjigeorgiou GM, Karatzaferi C, Maridaki MD, Koutedakis Y, Founta P, Tsianas N, Stefanidis I, Sakkas GK. A single-blind randomized controlled trial to evaluate the effect of 6 months of progressive aerobic exercise training in patients with uraemic restless legs syndrome. Nephrol Dial Transplant. 2013 Nov;28(11):2834-40. doi: 10.1093/ndt/gft288. Epub 2013 Aug 8. PMID 23929523